CLINICAL TRIAL: NCT05997888
Title: Examining the Feasibility, Acceptability, and Preliminary Efficacy of a Six-week At-home Strength Training Intervention for Black Women
Brief Title: Feasibility, Acceptability, and Preliminary Efficacy of a Six-week Physical Activity Intervention for Black Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Principal Investigator, Beth Lewis, Principal Investigator, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00019542
Record Dates: First submitted 2023-07-31; First posted 2023-08-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At-Home Strength Training Group (Experimental): Participants in this arm will undergo an in-person meeting before the start of the study to meet each other, go over movements to minimize risk of injury, and to discuss intervention logistics. Then, for six weeks, participants will be sent five workouts at the start of each week (Monday). Participants will choose 2 or 3 to complete on their own. Additionally, participants will have a weekly Zoom meeting in which 30 minutes will be dedicated to exercising, and 30 minutes will be for group counseling.
  Interventions: Behavioral: At-Home Strength Training Intervention
- Wait-List Control Group (No Intervention): This will be a wait-list control group. Participants at the end of the study will have the option to complete the full, partial, or none of the intervention.

INTERVENTIONS:
Behavioral: At-Home Strength Training Intervention — A six-week strength training intervention in which participants will choose workouts to complete on their own. These workouts are 20-25 minutes light-intensity strength training with light strength bands. Exercises will have multiple options to account for various levels of ability. Additionally, there will be a group counseling session once per week via Zoom and a group strength training program.
  Arms: At-Home Strength Training Group

SUMMARY:
The current study will be a randomized controlled pilot study conducted in the Midwest. Participants will be randomly assigned to a behavioral intervention or a wait-list control group, each lasting six weeks. The intervention group will first have an in-person meeting at the beginning of the intervention to discuss the study, go over movements, and discuss Zoom and WhatsApp instructions. The behavioral intervention will consist of three home-based workouts per week sent digitally and Zoom session per week that will have an exercise session and a group counseling session. Additionally, each week participants will be sent a motivational prompt via WhatsApp and will be encouraged to connect with each other about physical activity motivation, barriers, and facilitators. Acceptability, physical activity and psychosocial variables of interest will be measured via accelerometer data (via Actigraph GT3X) and self-report at baseline and six weeks (post-intervention). Focus groups will be conducted for all participants at the conclusion of the study to further assess acceptability, feasibility, and efficacy of the program.

DETAILED DESCRIPTION:
Step 1- Formative Focus Groups: Prior to recruitment of participants, three focus groups with five to eight members of the target population per group will be conducted to accomplish the following: 1) Review intervention materials such as exercise session content, motivational construct activities, and counseling session topics, and 2) assess any barriers and facilitators within their environments that should be accounted for in the methodology of the study, and 3) to explore how racism impacts their lives and how their ability to engage in physical activity. A trained consultant will ask questions regarding length of workouts, frequency of messaging on WhatsApp, whether video calls between participants and the PI would be helpful, and what type of messaging and video content the participants may like to see, in accordance with similar literature in the field (Joseph et al., 2017). Formative research participants will be paid $20 for their time. After the focus groups conclude, the PI and another researcher will conduct inductive hierarchical content analysis to incorporate results into the intervention structure and design. Audio and/or video recordings will be taken in order to accurately analyze themes and adjust the protocol based on answers from the focus groups. The protocol of the intervention will be adjusted with results from the formative focus groups after receiving relevant input.

Step 2- Telephone Screening, Consent, and Baseline Questionnaires: In response to advertisement and outreach efforts, potential participants will call, email, or text the Student Investigator (SI), at which time they will complete a telephone screening interview with the SI to determine eligibility for the study. Participants who are eligible will be given detailed information about the study and the consent form will be reviewed. The SI will schedule a randomization appointment in two weeks. Participants will be told that they may need to cancel the appointment if the online consent and questionnaires are not completed.

a) Complete telephone screening

1. If not eligible, end interview and thank them for their time
2. If eligible:

i. Schedule randomization appointment for 2 weeks ii. Email link to consent form and questionnaires iii. Explain ActiGraph procedures. The Actigraph is a small device that is attached to the participant's clothing/belt at the waist and measures physical activity amount and intensity. The Actigraph functions as a method of measuring physical activity with the purpose of obtaining objective measurement of the participants' physical activity.

Step 3- Send Actigraph: Upon completion of the consent form and questionnaires, send the Actigraph assessment with instructions and return envelope.

Step 4- Check on consent and baseline questionnaires: If the ActiGraph is not received by the randomization appointment, the participant is to be called to cancel the appointment. The participant should be told that they will be called to reschedule the appointment once the ActiGraph is received.

1. Once the ActiGraph is received, call the participant to schedule a time or if time permits, complete the randomization appointment at the time of the initial call.
2. If the ActiGraph has been received, proceed with the scheduled randomization appointment.

Step 5- Baseline Session:

1) Participants are randomly assigned to either the exercise or wait-list control condition. The wait-list control condition will have the option of receiving the exercise intervention after the 6 weeks. The exercise intervention will be delivered via phone. Enter randomization date in REDcap.

1. Script: "The next thing we are going to do is to find out which of the two groups you have been randomly assigned to. This is completely random and unfortunately I have no control over which group you are assigned to. Let me access my form here to determine which program you are in."
2. Exercise: "You have been randomly assigned to the exercise program. This program is designed to help you increase your exercise. I will work with you to make a plan on how you are going to fit exercise into your day. Do you have any questions before we start?"
3. Wait-List Control: "You have been randomly assigned to the wait-list control condition. This means that you will be contacted again in 6 weeks to complete your assessment. After your assessment, you will complete the exercise program if you would like to."

Step 6- Intervention Sessions (separate protocol is attached to submission):

1. The participant will be told when exercise should be stopped for safety reasons in order to minimize risk to the participant.
2. Baseline fitness will be assessed with a sit up and push up test (to assess strength and endurance) prior to the first meeting (this will be scheduled).
3. Participants randomly assigned to the behavioral intervention will begin with a 90 minute in-person meeting at a community space with all intervention participants, the SI, and the trained research assistant. At this meeting, participants will have time to meet each other and the researchers, and refreshments will be provided by the research team. The research team will show all participants how to download WhatsApp and join the group chat. Participants will also be instructed to use their first name only in the WhatsApp group chat in order to maintain confidentiality. Then, proper form for common movements that will be used in the intervention, such as squats, lunges, push-ups, and exercises with bands will be demonstrated and practiced by all participants. While participants practice these movements, the research team will provide feedback on exercise form to ensure that participants are using safe and proper techniques to avoid injury. Additionally, participants will receive information regarding the benefits of physical activity for physical and mental health, and will be encouraged to ask any questions they may have about the intervention or physical activity for health. Finally, all participants will be asked if they have any questions, and the PI will facilitate any questions and discussion during this time.
4. On Monday of each week, participants will be sent five workouts per week (depending on results from the focus groups) to their emails. All workouts will vary by time, number of exercises, and muscle group focus, but all involve bodyweight and banded strength exercises designed to be low intensity. Variations will be provided, and participants will be free to choose the variation that fits their comfortability level (e.g. push-up versus knee push-up). All workouts will slightly increase in difficulty each week in regard to repetition numbers and workout length but will have similar movements and structure. Workouts will either be targeted toward a specific muscle group or various muscle groups will be combined into one session. Of the five workouts sent per week, participants will be asked to complete two in the first half of the intervention (weeks one through three) and three in the second half of the intervention (weeks four through six).
5. Participants will be sent short motivational prompts via WhatApp (depending on results from the focus groups) on Monday of each week that target constructs of self-efficacy and motivation, as informed by Self-Efficacy Theory and Self-Determination Theory. Participants will be encouraged to respond to the prompt in the group and chat with each other as much as they want during each week. The SI will not participate in the group beyond sending a motivational prompt each week, and any questions for the PI will be answered via email so as not to interrupt the flow of engagement between participants. On each Monday, participants will also be instructed to send the SI which workouts they completed and on which days of the week.
6. Participants in the intervention group will engage in one 60-minute Zoom session per week to foster connectivity between participants and the research team. In the first 25 minutes, participants will engage in group counseling based on the motivational prompts sent out on Monday. After the counseling session, participants will then engage a 25-minute group exercise session that is similar to the sample workouts in regard to difficulty. Before the start of the exercise session, participants will be told to stop exercising if they experience shortness of breath, chest pain, and/or pain radiating down one arm, dizziness, muscle weakness, calf pain, or a headache. The first five minutes will be dedicated to stretching and warming up. The exercise session will last approximately 25 minutes, with twenty minutes for the main exercise session and five minutes will be a cool down and debrief of the session. During the exercise portion of the meeting, all participants will complete the Feeling Scale (FS) to assess feelings at different points of the exercise session. In the group counseling sessions, participants will engage in activities related to motivation for physical activity and they will work together to discuss how to overcome barriers to physical activity.

Step 7- 6-week assessment:

1. At 5 weeks, the participant will be mailed to the ActiGraph, which will be worn for one week starting the day after the last intervention session.
2. At 6 weeks, the participant will be prompted to complete the 6-week questionnaire.
3. The participant will be sent a $50 gift card once the assessment is complete and the ActiGraph is received.

Step 8- Post-Intervention Focus Group

1) At the conclusion of the intervention, the intervention group will undergo a one-hour focus group that will ask various questions regarding the intervention. These focus groups may be audio and/or video recorded (questions attached to submission)

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black
* Be categorized as insufficiently active, defined as less than 90 minutes of physical activity and less than two days of strength training
* Live in the Twin Cities area
* Be at least 18 years-old
* Be able to participate in the study for six weeks and agree to participate in a focus group at the conclusion of the study
* Possess a smartphone
* Be willing to wear an accelerometer (Actigraph GT3X) for the duration of the study
* Be able to attend a weekly 60 minute Zoom session on one of two selected nights
* Be willing to be randomized to the intervention or control condition.

Exclusion Criteria:

* Do not identify as Black
* Are active over 90 minutes per week
* Are under 18 years-old
* Will be unable to participate in the full study
* Do not possess a smartphone
* Are unwilling to wear an accelerometer
* Are unwilling to be randomized to either condition
* Are pregnant
* Have a serious physical or mental condition that would interfere with the ability to do physical activity
* Are currently enrolled in another exercise-related study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as a woman
Enrollment: 36 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of the programs | Six weeks
  Customer satisfaction. Feasibility of the intervention will be measured by looking at acceptability and implementation of the intervention. Level of acceptability will be assessed by examining the percentage of Zoom sessions (both group and individual) attended and self-reported number of exercise sessions completed per week. This measure will be assessed on a 1-7 point Likert scale, with one = "very dissatisfied" to seven = "very satisfied". Participants will be asked to rate their satisfaction on a variety of elements such as Zoom sessions, weekly WhatsApp messages, and the overall program.
Acceptability | Six weeks
  Acceptability will also be assessed with a customer satisfaction form, which asks participants to respond on a seven-point Likert scale, with one = "very dissatisfied" to seven = "very satisfied". Participants will be asked to rate their satisfaction on a variety of elements such as Zoom sessions, weekly WhatsApp messages, and the overall program.

SECONDARY OUTCOMES:
Social support | six weeks
  Physical Activity Social Support (PASS). The PASS scale is a 13-item measure that assesses family and peer support for physical activity within the past month. PASS asks respondents to gauge support with statements such as "did physical activity with me" and "criticized or made fun of me for doing physical activities" on a 5-point Likert scale ranging from 0 (none) to 4 (very often). The PASS has shown empirical validity and high test-retest reliability. Additionally, the PASS has had internal consistency scores ranging from ɑ = 0.61 to ɑ = 0.84.
Behavioral regulation | six weeks
  The Behavioral Regulation in Exercise Scale (BREQ-2, Markland & Tobin, 2004) was built off of Deci & Ryan's (2000) Self-Determination Theory to assess motivation for physical activity. The BREQ-2 consists of 19 items that ask why respondents exercise and assess motivation along a self-determination continuum of amotivation, external motivation, introjection, identification, integration, and intrinsic regulation. Respondents are asked whether statements on a scale of one ("not true for me") to four ("very true for me"). Internal consistency was above the standard for the field, ɑ = 0.749-0.849. The BREQ-2 has demonstrated sufficient reliability and validity.
Enjoyment | six weeks
  Physical Activity Enjoyment Scale (PACES). The Physical Activity Enjoyment Scale (PACES) is an 18-item measure to assess perceptions of physical activity. PACES asks respondents to "rate how you feel at the moment about a physical activity you have been doing." PACES uses a 7-point Likert scale and asks participants to respond to paired statements such as, "I am very absorbed in this activity" versus "I am not at all absorbed in this activity" and "It's very gratifying" versus "It's not at all gratifying." Eleven of the 18 items are reverse scored. PACES has demonstrated high internal consistency, ɑ = 0.93, and reliability. The PACES has demonstrated reliability and validity for various adult populations.
outcome expectations | six weeks
  Outcome Expectations for Exercise Scale (OEE). Outcome expectations, or the assessment of the consequences of a behavior, was gauged with the 9-item Outcome Expectations for Exercise Scale (OEES). OEE is based on Social Cognitive Theory, which postulates that outcome expectations influence physical activity behavior. Five items assess the physical benefits of exercise and four assess the mental benefits of exercise. Respondents are asked to read statements regarding perceived consequences of exercising and indicate on a five-item Likert scale whether they one (strongly agree) to five (strongly disagree). Items include statements such as exercising "makes me feel better physically" and "improves my endurance in performing my daily activities." The OEE has high internal consistency, ɑ = 0.95, and has been shown to have good validity and reliability in samples similar to the current study.
self-efficacy | six weeks
  Self-Efficacy. Self-efficacy for exercise will be assessed using a 5-item measure that asks participants to rate their confidence that they will be able to be physically active in five different situations (vacation, being tired, being busy, being in a bad mood, and inclement weather). This five-item likert scale varies from one = "not at all confident" to five = "extremely confident" (Marcus et al., 1992). This measure of self-efficacy has been validated for adult populations and has an internal consistency of ɑ = 0.76.
Physical Activity | six weeks
  The Actigraph GT3X has been empirically validated to objectively measure physical activity for adults. Accelerometers have provided empirically validated data and overcome many problems associated with self-report data, such as overestimation of physical activity. 7-Day PAR - This measure asks the participant to recall the amount of time for each day in the past seven days that they engaged in moderate, hard, and very hard physical activity. This measure has also shown moderate consistency when compared to accelerometer data.

OTHER OUTCOMES:
Themes from focus groups | six weeks
  Intervention participants will complete a focus group in which we ask various questions surrounding the intervention
Everyday discrimination | baseline
  The Everyday Discrimination Scale (EDS) is one of the most widely used measures in health research, and captures discrimination across various social groups, including race, gender, and weight. Participants are asked to indicate frequency surrounding experiences in their day-to-day lives, such as "You are treated with less courtesy than other people are", or "People act as if they are afraid of you." The EDS is scored on a six-point Likert scale, with a 0 = "Never" and a 5 = "Almost everyday." Then, to those participants who responded with at least "A few times per year" to any of the original questions are then asked "what do you think is the main reason for these experiences?" The EDS has reported an internal consistency of ɑ = 0.80-0.88, and sufficient construct, predictive, and convergent validity.
Hair type and hairstyle management | baseline and six weeks
  The Hair Type and Hairstyle Management (HTHM) scale was developed in order to understand hair care and hairstyle for Black women to assess hair as a potential obstacle for physical activity for Black women. This measure asks questions regarding natural hair structure, use of chemical treatment or relaxers, current hairstyle, average cost per month of hair care, and whether participants alter behavior due to hair concerns.
Feeling Scale | weekly (weeks 2-6)
  intervention participants will take this measure every Zoom counseling session, three times per session to assess how they're feeling and how much they're enjoying the exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No